CLINICAL TRIAL: NCT00456924
Title: Prospective Randomized Multicenter Phase II Study of the Dose-Response Effects of Continuous Administration of Low-Dose VA2914 on Parameters of the Hypothalamic-Pituitary-Gonadal Axis and the Endometrium
Brief Title: Low Dose Continuous Administration of the Progesterone Receptor Modulator VA2914
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2914-002
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Contraception; Gynecologic Diseases
Keywords: progesterone receptor modulator
MeSH Terms: conditions — Genital Diseases, Female | interventions — ulipristal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: VA2914

SUMMARY:
The purpose of the present study is to evaluate continuous administration of low doses of VA2914 for potential contraceptive activity and effects on the menstrual cycle and steroid hormone parameters.

ELIGIBILITY:
Inclusion Criteria:

* women in good general health with regular, ovulatory menstrual cycles
* age 18-35
* not pregnant
* not sexually active or reliably use barrier methods of contraception
* normal liver and renal functions and normal laboratory exams

Exclusion Criteria:

* pregnant or breastfeeding
* oral contraception, IUD or other hormonal treatment
* use of agents known to induce hepatic P450
* cardiovascular disorder
* hepatic, renal, or gastrointestinal disorder
* metrorrhagia
* abnormal transvaginal ultrasound (at baseline)
* history of abnormal endometrial biopsy,
* cancer
* depression
* mental illness
* epilepsy
* migraines
* abnormal Pap Smear requiring further exploratory examination
* anovulatory cycle before treatment
* extreme overweight or underweight (body mass index < 16 ou >28)
* subjects unlikely to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* use of narcotics
* more than 10 cigarettes per day, more than 2 glasses of wine/beer per day
* surgical procedures planned in the 6 months following screening visit

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48
Dates: Start 2004-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
ovarian hormones
follicular development
endometrial histology

SECONDARY OUTCOMES:
menstural bleeding patterns
cervical mucus
VA2914 concentration
adverse events
laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bouchard, MD, Principal Investigator — Saint Antoine Hospital, Paris, France
Locations (4):
- Belgium (2):
  - Liege University Hospital, Liège
  - Sainte Rosalie Clinique, Liège
- France (2):
  - Antoine Beclere Hospital, Clamart
  - Saint Antoine Hospital, Paris

REFERENCES:
- [Result] Chabbert-Buffet N, Pintiaux-Kairis A, Bouchard P; VA2914 Study Group. Effects of the progesterone receptor modulator VA2914 in a continuous low dose on the hypothalamic-pituitary-ovarian axis and endometrium in normal women: a prospective, randomized, placebo-controlled trial. J Clin Endocrinol Metab. 2007 Sep;92(9):3582-9. doi: 10.1210/jc.2006-2816. Epub 2007 Jun 19. PMID 17579200